CLINICAL TRIAL: NCT04830852
Title: Pediatric SARS-CoV-2 and MIS-C Long-term Follow-up
Brief Title: Pediatric COVID Outcomes Study (PECOS)
Status: Active, not recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Roberta DeBiasi, MD, MS, Division Chief, Infectious Diseases, Co-Director of the Congenital Zika Program, Children's National Research Institute
Other Study IDs: Pro00015510; 21X125F1 (Other: Leidos)
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: Covid19; MIS-C Associated with COVID-19; MIS-C Multisystem Inflammatory Syndrome in Children; SARS-CoV2 Infection
Keywords: SARS-CoV-2; COVID-19; MIS-C; Post-COVID; Long-term effects; Pediatric; Children
MeSH Terms: conditions — COVID-19; pediatric multisystem inflammatory disease, COVID-19 related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, nasopharyngeal swab, stool and urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Recovery Group: Participants aged 21 years and younger and enrolled within 12 weeks after acute infection or positive test. These participants will attend study visits at baseline, every 3 months for the first 6 months, and subsequently every 6 months for a total of 3 years.
- Convalescent Group: Participants aged 21 years and younger and enrolled more than 12 weeks after acute infection or positive test. These participants will attend study visits at baseline and subsequently every 6 months for a total of 3 years.
- Healthy contacts: Individuals (aged ≤21 years) without a diagnosis of SARS-CoV-2 infection or current symptoms suggestive of COVID-19 will serve as a control group and will attend visits for evaluations and sample collection at baseline and every 12 months for a total of 3 years.
- Parents/guardians of participants: Parents or guardians of participants in all cohorts will also be enrolled for limited participation to complete questionnaires about how the family is impacted by the participant's health and SARS-CoV-2.

SUMMARY:
This is a multisite prospective observational study to evaluate the clinical sequelae of symptomatic and asymptomatic severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection in the pediatric population, including coronavirus disease 2019 (COVID-19) and multisystem inflammatory syndrome in children (MIS-C), and characterize the immune response associated with these clinical presentations. Participants aged 21 years and younger with laboratory confirmed history of symptomatic or asymptomatic SARS-CoV-2 infection will visit the study sites for clinical and research evaluations and sample collection at schedules dependent on time since infection. Participants enrolled within 12 weeks after acute infection or positive test will be part of the "recovery group" and will attend study visits at baseline, every 3 months for the first 6 months, and subsequently every 6 months for a total of 3 years. Participants enrolled more than 12 weeks after acute infection or positive test will be in the "convalescent group" and will attend study visits at baseline and subsequently every 6 months for a total of 3 years.

Individuals (aged ≤21 years) without a diagnosis of SARS-CoV-2 infection or current symptoms suggestive of COVID-19 will serve as a control group and will attend visits for evaluations and sample collection at baseline and every 12 months for a total of 3 years. This protocol will establish a cohort of pediatric patients recovered from SARS CoV-2 infection and a biorepository for evaluation of the potential roles of host genetics, immune response, and other possible factors influencing long-term outcomes.

Parents or guardians of participants in all cohorts will also be enrolled for limited participation to complete questionnaires about how the family is impacted by the participant's health and SARS-CoV-2.

DETAILED DESCRIPTION:
This study will establish a cohort of surviving pediatric patients with symptomatic (including COVID-19 and MIS-C) and asymptomatic SARS-CoV-2 infection to study the long-term sequelae of acute infection and the evolution of the immune response over time. Longitudinal follow-up of this cohort will provide important information about clinical sequelae of acute COVID-19 and MIS-C, characteristics of the immune response to SARS-CoV-2, genetic factors associated with long-term outcomes, and the extent and duration of protective immunity.

The study procedures include:

1. Non-contrast chest computed tomography (CT) or chest X-ray: All participants will undergo 2 chest imaging procedures, one at baseline and one at the final study visit (year 3).
2. Non-contrast cardiac magnetic resonance imaging (MRI): All participants will undergo 2 to 3 non-contrast cardiac MRI procedures during this study.
3. Echocardiogram
4. Electrocardiography (EKG)
5. Pulmonary Function Test (PFT)
6. Questionnaires: To complete the questionnaires will take approximately 25 to 64 minutes.
7. Collection of blood (including for optional genetic testing), nasopharyngeal (NP) swab, urine, and stool.

Genetic testing (optional): This protocol involves genetic testing using whole genome sequencing (WGS) approaches for all participants.

Clinical photography (optional): Participants may decline photographs or place any restrictions on their use.

ELIGIBILITY:
Inclusion Criteria:

Survivors and control cohorts:

In order to be eligible to participate in this study as a survivor or as a control, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Male or female aged 0 to 21 years (at the NIH CC, minimum age is 3 years).
3. Willing to allow storage of samples and data for future research.
4. At the NIH CC: Has a physician or clinic outside NIH to manage underlying medical conditions, or agrees to establish care with an outside physician or clinic for any medical conditions requiring treatment that may be diagnosed as a result of protocol participation.

In addition, an individual must meet all criteria for one of the following cohorts.

Symptomatic survivor cohort (including MIS-C):

1. Documented prior COVID-19 or MIS-C as evidenced by one of the following:

   1. detection of SARS-CoV-2 RNA or antigen in NP swab, saliva, sputum, or other sample source with Emergency Use Authorization (EUA)/approval from the US Food and Drug Administration (FDA) and a history of clinical manifestation compatible with COVID-19*; or
   2. positive SARS-CoV-2 antibody test using an assay that has received EUA from the FDA (negative SARS-CoV-2 RNA or antigen or never tested), and a history of clinical manifestation compatible with COVID-19*; or
   3. meeting CDC case definition for MIS-C (see Appendix 1).
2. Onset of COVID-19/MIS-C symptoms is at least 4 weeks before baseline visit. *one or more of the following: ageusia, anosmia, chills, confusion, cough, rash, "COVID toes", diarrhea, dyspnea, fatigue, fever, headache, myalgia, nausea/vomiting, pneumonia, rhinorrhea.

Asymptomatic survivor cohort:

1. Documented prior SARS-CoV-2 infection as evidenced by one of the following:

   1. detection of SARS-CoV-2 RNA or antigen in NP swab, saliva, sputum, or other sample source with EUA/approval from the FDA without history of clinical manifestation compatible with COVID-19; or
   2. positive SARS-CoV-2 antibody test using an assay that has received EUA from the FDA without history of clinical manifestation compatible with COVID-19*.
2. Positive SARS-CoV-2 RNA or antigen test is at least 4 weeks before baseline visit.

   * one or more of the following: ageusia, anosmia, chills, confusion, cough, rash, "COVID toes", diarrhea, dyspnea, fatigue, fever, headache, myalgia, nausea/vomiting, pneumonia, rhinorrhea.

Healthy contact (control) cohort:

1. No diagnosis of SARS-CoV-2 infection or current symptoms suggestive of COVID-19 and meets one of the following criteria:

1. Lived in the same household as a participant with SARS-CoV-2 infection during the time of illness, or was within approximately 6 feet (2 meters) of the participant for a prolonged period of time, or having direct contact with infectious secretions of a COVID-19 case (e.g., being coughed on).
2. Lives in an area affected by SARS-CoV-2 infection

Parents and guardians:

In order to participate in this study as a parent or guardian, an individual must meet all of the following criteria:

1. Is a parent or guardian of a participant enrolled as a survivor or as a control.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Willing to allow storage of data for future research.

Exclusion Criteria:

Survivors and controls:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any symptoms suggestive of an ongoing infection within 15 days of baseline visit, including but not limited to fever > 38.2 °C, new or worsening respiratory symptoms (e.g., cough, dyspnea), or new or worsening gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea or abdominal pain).
2. Any medical or mental health condition that, in the judgement of the principal investigator, would make the volunteer unable to participate in the study.
3. Pregnancy.

Parents and guardians:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any medical or mental health condition that, in the judgement of the principal investigator, would make the volunteer unable to participate in the study.

Co-enrollment: Participants may be co-enrolled in other clinical studies, including observational studies and therapeutic trials. However, the study staff should be informed of co-enrollment.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients aged 0 to 21 years with confirmed history of symptomatic SARS CoV-2 infection (including COVID-19), MIS C, or asymptomatic SARS CoV-2 infection (n = up to 1000), as well as healthy contacts (aged ≤21 years; n = up to 1000). Additionally, a parent or guardian of each participant will be enrolled to complete targeted questionnaires (n = up to 2000).
  Accrual ceiling is 5000 patients.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and prevalence of medical sequelae, study procedures analysis | 6 years
  Incidence and prevalence of medical sequelae among symptomatic SARS-CoV-2 infection survivors, asymptomatic SARS CoV 2 infection survivors, and MIS-C survivors.
Risk factors for medical sequelae, study procedures analysis | 6 years
  Risk factors for medical sequelae among symptomatic SARS CoV 2 infection survivors, asymptomatic SARS-CoV-2 infection survivors, and MIS-C survivors.

SECONDARY OUTCOMES:
Quality of life and social impact, study procedures analysis | 6 years
  Health-related quality of life and social impact in children and adolescents recovered from SARS-CoV-2 infection including parent/guardian and child assessments.
Incidence and prevalence of reinfection, study procedures analysis | 6 years
  Incidence and prevalence of reinfection in previously infected and recovered SARS-CoV-2 and MIS-C survivors with and without vaccination.
Biorepository, study procedures analysis | 6 years
  Establishment of a biorepository for additional biomarker analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta DeBiasi, MD, MS, Principal Investigator — Children's National Research Institute; Gina A. Montealegre Sanchez, MD, MS, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - Children's National Hospital, Washington D.C., District of Columbia
  - National Institutes of Health (NIH) / National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland

REFERENCES:
- See also: If you are interested in participating in this study, please complete this form. A study team member will contact you with additional information. — https://childrensnational.formstack.com/forms/covid_misc_study